CLINICAL TRIAL: NCT05185206
Title: Comparative Evaluation of the Post Operative Sensitivity of Cention-N(Commercially Available Restorative Material) Using Conventional and Polymer Bur- In-vivo Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. D. Y. Patil Dental College & Hospital (Other)
Responsible Party: Principal Investigator, Soumya Shetty, Professor, Dr. D. Y. Patil Dental College & Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DYPDCH/IEC/123/99/19
Record Dates: First submitted 2021-12-12; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Dental Caries; Dentin Sensitivity
MeSH Terms: conditions — Dental Caries; Dentin Sensitivity

STUDY DESIGN:
Intervention Model Description: A split mouth study design which checks the post operative sensitivity with cention-n(commercially available restorative material) using conventional steel bur and polymer bur using Visual Analog scale.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants, investigator and outcome assessor will be blinded to the treatment modalities.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Analysis of post-operative sensitivity after caries removal using conventional steel bur (Active Comparator): Caries will be excavated using a carbide on one side of the arch and restoration will be done with Cention-N(commercially available restorative material) as per manufacturer's instructions.Thermal stimulation (refrigerant spray Endo-Ice) will be used to evaluate the type of sensitivity. The pain intensity will be recorded with the Visual Analog Scale.
  Interventions: Device: Class 1 cavity preparation using conventional steel bur and restoration with Cention-n(commercially available restorative material).
- Analysis of post-operative sensitivity after caries removal using polymer bur (Experimental): Caries will be excavated using a polymer on one side of the arch and restoration will be done with Cention-N(commercially available restorative material) as per manufacturer's instructions.Thermal stimulation (refrigerant spray Endo-Ice) will be used to evaluate the type of sensitivity. The pain intensity will be recorded with the Visual Analog Scale.
  Interventions: Device: Class 1 cavity preparation using polymer bur and restoration with Cention-n(commercially available restorative material).

INTERVENTIONS:
Device: Class 1 cavity preparation using conventional steel bur and restoration with Cention-n(commercially available restorative material). — Patients aged between 18 and 55 years having class 1 occlusal caries(1.2 according to G. J. Mount classification) on both sides of arch. In order to standardise the cavity preparation depth(approximately 1.5 to 2mm from the roof of the pulp chamber), the distance from occlusal surface to roof of pulp chamber will be used for measuring with the radiograph. This will be followed by caries removal with convention steel bur followed by restoration with Cention-n and checking of postoperative sensitivity using Visual Analog Scale.The Visual Analog Scale consists of a 100-mm line divided into equal intervals of 10 mm, where 0 represents "absence of pain" and 100 "severe pain." The results of Visual Analog Scale will be classified as mild (0-30 mm), moderate (40-70 mm), or severe pain (> 70 mm).
  Arms: Analysis of post-operative sensitivity after caries removal using conventional steel bur
Device: Class 1 cavity preparation using polymer bur and restoration with Cention-n(commercially available restorative material). — Patients aged between 18 and 55 years having class 1 occlusal caries(1.2 according to G. J. Mount classification) on both sides of arch. In order to standardise the cavity preparation depth(approximately 1.5 to 2mm from the roof of the pulp chamber), the distance from occlusal surface to roof of pulp chamber will be used for measuring with the radiograph. This will be followed by caries removal with polymer bur followed by restoration with Cention-n and checking of postoperative sensitivity using Visual Analog scale.The Visual Analog Scale consists of a 100-mm line divided into equal intervals of 10 mm, where 0 represents "absence of pain" and 100 "severe pain." The results of Visual Analog Scale will be classified as mild (0-30 mm), moderate (40-70 mm), or severe pain (> 70 mm).
  Arms: Analysis of post-operative sensitivity after caries removal using polymer bur

SUMMARY:
Cention-N(commercially available restorative material) is a cost effective restoration for posterior restorations. Post-operative sensitivity is of great concern as far as any type of restorative material is concerned. Reduction of post-operative sensitivity is still a major on-going research. Timely advancement has lead to the discovery and usage of polymer bur for reduction of excess tooth removal, and thus reduction of sensitivity. Therefore the novelty of this study is comparision of the post operative sensitivity of Cention-N(commercially available restorative material) using conventional and polymer bur using Visual Analog Scale.

DETAILED DESCRIPTION:
Dental caries is a multifactorial disease which is very much prevalent in India occurring especially in high economic group and some in middle and lower economic groups of world population.The most common instruments used for excavation of dental caries are the use of diamond and carbide burs.There is effective removal of the carious tooth structure through these burs which leads to excess removal of tooth structure and weakening the teeth.

Timely advancement in dentistry and the quest for the development of ideal esthetic materials to replace lost dental tissue has led to use of Cention-N(commercially available restorative material) to restore posterior teeth. Cention N(commerically available restorative material) is a recently introduced tooth-coloured, basic filling material for bulk placement in retentive preparations with or without the application of an adhesive. It is an alkise restorative which is a new category of filling material, like compomer(commercially available restorative material) or ormocer(commercially available restorative material) and is essentially a subgroup of the composite resin. Cention-N(commercially available restorative material)offers a cost-effective substitute for amalgam and also fulfills the need of an esthetic bulk fill material in the posterior region. Patients have described post-operative sensitivity as a moderate pain, of short duration, that appears spontaneously when chewing, with hot and cold foods and on rare occasions with sweet and acid foods, and it disappears when the stimulus is removed. It is characterized by an acute pain that can last for days or weeks and disappears when the stimulus is removed.It results from the interaction between the restorative technique, the clinical condition of the tooth to be treated (health of the pulp and remaining hard dental tissue) and the restorative material. Therefore, there is a permanent and unpredictable possibility of sensitivity occurring. In addition, there are other factors related to the cause of post- operative sensitivity, such as the individual profile of each patient, the shape and extension of the cavity preparation and protection of the dentin-pulp complex. Hence the novelty of this study is to evaluate of the post operative sensitivity of Cention-n (commerically available restorative material)using conventional and polymer bur.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 55 years having class 1 occlusal caries(1.2 according to G. J. Mount classification) on both sides of arch. In order to standardise the cavity preparation depth(approximately 1.5 to 2mm from the roof of the pulp chamber), the distance from occlusal surface to roof of pulp chamber will be used for measuring with the radiograph.
* Roots with closed apex.
* Systematically healthy patients.
* Patients with no other symptomatic tooth involved

Exclusion Criteria:

* Teeth with the presence of any pathologic pulpal disease with or without pain.
* Teeth with previous restorations, any defective restoration adjacent to or opposing the affected tooth.
* Teeth with surface loss due to attrition, erosion, abrasion, or abfraction.
* Patients with poor oral hygiene, severe, or chronic periodontitis.
* Patient on medication which may hinder the response to sensitivity.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-05-02 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Post-operative sensitivity checked using Visual Analog Scale by thermal stimulus. | Post operative sensitivity will be checked after 24 hours.
  Thermal stimulation (refrigerant spray Endo-Ice) will be used to evaluate the type of sensitivity. The pain intensity will be recorded with the visual analog scale (VAS).
Post-operative sensitivity checked using Visual Analog Scale by thermal stimulus. | Post operative sensitivity will be checked after 15 days.
  Thermal stimulation (refrigerant spray Endo-Ice) will be used to evaluate the type of sensitivity. The pain intensity will be recorded with the visual analog scale (VAS).
Post-operative sensitivity checked using Visual Analog Scale by thermal stimulus. | Post operative sensitivity will be checked after 30 days.
  Thermal stimulation (refrigerant spray Endo-Ice) will be used to evaluate the type of sensitivity. The pain intensity will be recorded with the Visual Analog Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr D.Y. Patil Dental College and Hospital, Pimpri, Pune, Maharashtra, India